CLINICAL TRIAL: NCT04378517
Title: Evaluation of the Feasibility of Family Strength-oriented Therapy Conversation for Families of 13-18 Years Old Adolescents With Attention-Deficit/Hyperactivity Disorder, at the Child and Adolescent Outpatient Unit: A Pilot Study
Brief Title: Evaluating the Feasibility of FAM-SOTC Intervention for Families of Adolescents With ADHD: Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iceland (Other)
Responsible Party: Principal Investigator, Erla Kolbrún Svavarsdóttir, professor, University of Iceland
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UI-2019_ADHD-pilotstudy
Record Dates: First submitted 2020-05-04; First posted 2020-05-07 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Attention Deficit Hyperactivity Disorder Combined
Keywords: ADHD; adolescents; advanced psychiatric nursing; caregivers; family strength therapeutic conversation; psychosocial education; psychosocial support
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Interviews as Topic

STUDY DESIGN:
Intervention Model Description: Pilot-study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ADHD FAM-SOTC support: A Pilot Study (Other): Phase-I, a pilot study to evaluate the feasibility of offering a 5-week intervention for families of adolescents diagnosed with ADHD at BUGL. The outcome helps to determining the feasibility of subjecting the intervention to a more rigour and a more expensive and time-consuming RCT.
  Phase-II and III are an RCTs to determine the benefit of a FAM-SOTC intervention: Is there a significant difference in the impact of FAM-SOTC intervention:
  From caregiver's perspective (phase II) on the experience of support for, family functioning, believes, coping patterns, general well-being, parental adaptation and parental assessment of ADHD symptoms and adolescent developmental disruptive behaviour, compared to caregivers receiving delayed treatment?
  From adolescents' perspective (Phase-III) in the assessment of adolescents own self-awareness and self-esteem, after their parents receive FAM-SOTC intervention, compared to a group of adolescents where caregivers receive delayed treatment?
  Interventions: Other: psychosocial education in parents groups; Other: psychosocial parents support, interviews with APN

INTERVENTIONS:
Other: psychosocial education in parents groups — psychosocial education
Other: psychosocial parents support, interviews with APN — Family strength-oriented therapy conversation

SUMMARY:
Attention-deficit/hyperactivity disorder (ADHD), is a highly genetic and complex neurological disorder, where disruptive behavior, emotional imbalance, and lack of attention can interrupt with normal development of adolescents, self-awareness, and self-regulation in a way that has an impact on the family unit. Effective family intervention programs, that empower resilience and strength, to cope with the stressful situation from ADHD, are therefore needed. Nevertheless, there is a lack of knowledge regarding what type of interventions are the most effective for these families. As well as, little is known about the benefits of family-level intervention for families of adolescents with ADHD at outpatient care and what amount of combination in an intervention is appropriate. Psychiatric advanced practical nurse (APN) practitioners are in a key role to offer such an intervention. Therefore, the aim of this pilot study is to evaluate the feasibility of offering a family-level intervention, for parents of 13-17 years old adolescents with ADHD, at a Children and Adolescents' Psychiatric Outpatient Unit (BUGL). Also, to evaluate if the intervention, which consists of group educational sessions, family sessions, and access to evidence-based information's on ADHD, fitted the families.

A nurse-led educational and support intervention will be offered for parents of adolescents with ADHD once a week over a 5-week time period. First, there will be offered three group support sessions, with information about the general impact of the ADHD disorder on the family's daily life. Second, two special therapeutic conversations and support interviews will be offered to each family, where each parent can discuss their daily situation specifically and its impact on the family as a whole. Third, caregivers will have access to about 140 pages of evidence-based material on a closed website (pan pale) regarding the ADHD disorder in adolescents and its impact on the family.

The outcome of this process will help in determining the feasibility of subjecting the intervention to a more expensive and time-consuming randomized controlled trial (RCT) study.

DETAILED DESCRIPTION:
A pilot study is a cornerstone to represent many methodological design challenges when studying a vulnerable group of parents or when testing the feasibility of an intervention. Attrition of dropout is one of the most crucial components in intervention research for families of adolescents in third-line care as for families of adolescents with ADHD. Furthermore, motivation is important to keep parents engaged, as well as to minimize the risk of them dropping out of the study. In a pilot study, questions are asked regarding if the intervention can be done, and it is determined whether an intervention warrants further testing, and if so, how. This special design then elements the study as a small-scale study, before the main full-size study will be conducted. Further, this design of a study is also done to improve the quality, to evaluate the safety of the intervention, to re-evaluate the recruitment possibilities as well as to considering ethical aspects of a larger randomized control trial (RCT) study. This pilot study is therefore conducted to assess the feasibility of a 5-week Family strength-oriented therapy conversation (FAM-SOTC) intervention in an RCT. Preliminary research is used to assess the process, resources, management, and scientific value. This is an important factor in increasing the efficiency and results of future RCTs and preventing wasted time and resources.

From November 2018 until March 2019, will caregivers of adolescents aged 13-18 with a diagnosis of ADHD at BUGL be randomly selected and invited to participate in the study. Inclusion criteria for family participation are (a) adolescents diagnosed with ADHD at BUGL and (b) born between 2001 and 2007. (c) Caregivers needed to speak and read fluent Icelandic and (d) be living close to the capital city. Exclusion criteria are (a) caregivers not speaking or reading fluent Icelandic and (b) the family living in the countryside

The FAM-SOTC intervention emphasizes the family's strength and resilience, empowering parents of adolescents with ADHD to support themselves and their child. The FAM-SOTC requires nurses to build trust in the therapeutic relationship, listen to families, reflect on therapeutic questions, and offer appropriate evidence-based information and guidelines. The FAM-SOTC is based on the Calgary family assessment model (CFAM) and Calgary family intervention model (CFIM), as well as the illness beliefs model (IBM), which views suffering as stemming from the beliefs about the illness, but not the illness itself. Addressing beliefs about the illness presents a new path for helping families to handle stressful situations. In addition, Barkley's clinical manual for family assessment and intervention are used to guide caregivers step-by-step in how to deal with demanding ADHD symptoms. Clinical advice will be given to strengthen the supportive role of parents to improve the parent-teen relationship and the adolescent's adjustment.

The 5-week family strength-oriented therapeutic conversation intervention proceeded as follows: caregivers will be invited to participate once a week over a 5-week time period. First, a two-hour ADHD educational and psychosocial group support sessions will be held for caregivers (five families in a group, one per week over a 3-week period) that included general ADHD information, a 10-step process for supporting adolescents in a positive, constructive way, and problem-solving exercises to practice in the group and at home (a total of six hours of educational and psychosocial support sessions). Second, APNs led special therapeutic conversations and provided individualized support for each family (once a week for 2 weeks; 60-90 min each section, resulting in 2-3 hours of support for each family). The individualized support emerged from the therapeutic relationship and family relations and allowed caregivers to tell their narrative illness stories. Therapeutic questions are used for assessment (CFAM) of caregivers' strengths, resiliency, and resources to understand their need for further guidance and to recommend interventions (build on the CFIM) to identify facilitate and/or constrain beliefs. Thereby, the FAM-SOTC can strengthen family functioning, well-being, illness beliefs, and family support. Third, over the whole study period, parents received access to a website with about 140 pages of evidence-based (EB) - educational and informative material to be used as they wished.

At the beginning of the study, participants will provide written informed consent with agreeing to participate. Data will be collected with accurate, reliable questionnaires through the research electronic data capture (REDCap) data management platform. Caregivers and adolescents answer different questionnaires at the same time. The baseline measurement is taken at time one (t1) before caregivers received the intervention, and follow-up questionnaires are given at time two (t2) after the intervention (post-intervention), 5-weeks from baseline (t1).

The following instruments will be used for caregivers to measure their satisfaction and changes in their adolescents' ADHD symptoms: family-support (ICE-FPSQ); illness beliefs (ICE-FIBQ); family-activity (ICE-EFFQ); coping health inventory for parents (CHIP); the general well-being schedule (GWB); treatment evaluation questionnaire (TEQ); paediatric quality of life questionnaire (PedsQL); ADHD Rating Scale-IV (ADHD-RS); adolescents Disruptive Behaviour Rating Scale (DBRS); and background list in which information about gender, age, education, work, family status, diagnoses, and other psychological treatment are selected. The instruments for the adolescents to measure their self-esteem and mastery before and after their parents received the intervention are the Rosenberg Self-Esteem scale (50) and the Perlin et.al Mastery scale, in addition to a background questionnaire in which information about gender, age and education will be recorded.

Data analysis are based on Polit and Beck's implementation of descriptive statistics: 1) determine how many will agree to participate, 2) calculate median (the middle number) and interquartile range (IQR) (IQR = Q3-Q1, a measure of the spread of the number of sessions completed and mean length of time to complete the data collection form), 3) compute effect sizes and confidence intervals around estimates, 4) assess whether, for each person a reliable improvement will occur, 5) determine whether, a clinically significant change will occur in a responder analysis, 6) assess whether changes and benchmarks will be established to decide the feasibility, or if larger research is needed for the results to be deemed meaningful.

Ethic guidelines from the International Council of Nursing for ethical principles with human beings will be used. Before families agree to participate in the study, they receive an email with information about their role in the research, the nature of the study, and data collection. In addition, they will receive contact information from a psychiatrist, in case if they will experience discomfort with participating. Those that can not participate when invited have the opportunity to participate later and those that chose to receive the intervention but not answer the questionnaires will receive the intervention without participating in the study. Participating in the study has no effect on other treatment offered at the Psychiatric Unit; participants received the treatment as usual.

This feasibility study will help assess whether it is worth evaluating the 5-week FAM-SOTC intervention in a larger RCT study. As well as, representing methodological challenges for these families in a combination with a protocol of educational and support program for families of adolescents with ADHD to enhance adolescents' self-management behaviors. The results will be of interest to health care professionals working with ADHD adolescents patients. Additionally, our study will be of value to user organizations and policymakers administering education and support programs aimed at the prevention and treatment of ADHD in adolescents. In a way, to encouraging and empowering parents of adolescents wiht ADHD at psychiatric outpatient unit in their parenting caring role that can affect the families as a whole in a positive way.

ELIGIBILITY:
Inclusion Criteria: (a) Adolescents, aged 13-17 diagnosed with ADHD at a Children's and Adolescent's Psychiatric unit at Landspitali - The National University Hospital of Iceland (BUGL). (b) Born between 2001 and 2007. (c) Caregivers needed to speak and read fluent Icelandic and (d) be living close to the capital city.

Exclusion Criteria: (a) Caregivers do not speak or read fluent Icelandic and (b) the family live in the countryside.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 23 (Actual)
Dates: Start 2018-11-13 (Actual); Primary Completion 2019-02-20 (Actual); Study Completion 2019-03-27 (Actual)

PRIMARY OUTCOMES:
Iceland-Family Perceived Support Questionnaire (ICE- FPSQ). | T1 (at baseline in experimental group).
  The ICE-FPSQ is a 14-item questionnaire about support and education perceived from nurses within of two categories: cognitive and emotional support. It uses a scale with a scoring from 1-5; the higher scores indicate a better family function.
Iceland-Family Perceived Support Questionnaire (ICE- FPSQ). | T2 (post-intervention in experimental group, 6 weeks from T1)
  The ICE-FPSQ is a 14-item questionnaire about support and education perceived from nurses within of two categories: cognitive and emotional support. It uses a scale with a scoring from 1-5; the higher scores indicate a better family function.
Iceland-Family Illness Beliefs Questionnaire (ICE-FIBQ) | T1 (at baseline in experimental group).
  The ICE-FIBQ is a 7-item instrument that measure beliefs regarding illnesses among families who had members suffering from long-term illnesses. The questionnaire is a 5-point scale; higher scores indicate more reassurance regarding caregiver beliefs.
Iceland-Family Illness Beliefs Questionnaire (ICE-FIBQ). | T2 (post-intervention in experimental group, 6 weeks from T1).
  The ICE-FIBQ is a 7-item instrument that measure beliefs regarding illnesses among families who had members suffering from long-term illnesses. The questionnaire is a 5-point scale; higher scores indicate more reassurance regarding caregiver beliefs.
Iceland-Expressive Family Functioning Questionnaire (ICE-EFFQ). | T1 (at baseline in experimental group).
  ICE-EFFQ is a 17-item instrument within four categories: emotions, collaboration and problem-solving, communication and behavior. The questionnaire is a 5-point scale with a scoring range from 1 to 5; a higher score indicates a good family function.
Iceland-Expressive Family Functioning Questionnaire (ICE-EFFQ). | T2 (post-intervention in experimental group, 6 weeks after baseline).
  ICE-EFFQ is a 17-item instrument within four categories: emotions, collaboration and problem-solving, communication and behavior. The questionnaire is a 5-point scale with a scoring range from 1 to 5; a higher score indicates a good family function.
Treatment Evaluation Questionnaire | T2 (post-intervention in experimental group, 6 weeks after baseline).
  Caregivers answered a questionnaire regarding group care giving sessions and individual care giving sessions regarding education, conversation, tasks, and support. Answers to the questionnaire are either given as yes/no, open answers or a 5-point scale with a scoring range from 1 to 5; a higher score indicates a more positive experience.
Coping health inventory for parents (CHIP) | T1 (at baseline in experimental group).
  The CHIP measures parental coping patterns when parents have a child who is seriously and/or chronically ill. The CHIP comprises three sub-scales (dimensions) measuring three different coping patterns: a) maintaining family integration, co-operation, and an optimistic definition of the situation; b) maintaining social support, self-esteem, and psychological stability; and c) understanding the healthcare situation through communication with other parents and consultation with the healthcare team. The questionnaire is a 5-point scale; higher scores indicate more coping ability.
Coping health inventory for parents (CHIP) | T2 (post-intervention in experimental group, 6 weeks after baseline).
  The CHIP measures parental coping patterns when parents have a child who is seriously and/or chronically ill. The CHIP comprises three sub-scales (dimensions) measuring three different coping patterns: a) maintaining family integration, co-operation, and an optimistic definition of the situation; b) maintaining social support, self-esteem, and psychological stability; and c) understanding the healthcare situation through communication with other parents and consultation with the healthcare team. The questionnaire is a 5-point scale; higher scores indicate more coping ability.
The General Well-Being Schedule (GWBS) | T1 (at baseline in experimental group).
  GWBS is an 18-item instrument measuring positive and negative feelings: anxiety, depression, general health, positive well-being, self-control and vitality. The first 14 questions are 6-point scale (1=all of the time, 6=none of the time) and questions 15-18 are 1-10-point rating scales defined by adjectives feeling at each end.
The General Well-Being Schedule (GWBS) | T2 (post-intervention in experimental group, 6 weeks after baseline).
  GWBS is an 18-item instrument measuring positive and negative feelings: anxiety, depression, general health, positive well-being, self-control and vitality. The first 14 questions are 6-point scale (1=all of the time, 6=none of the time) and questions 15-18 are 1-10-point rating scales defined by adjectives feeling at each end.
The PedsQL-Family Impact Module. | T1 (at baseline in experimental group).
  The Family Impact Module is an instrument of 37 items that measures family's quality of life. Eight sub-scales of parents functioning that compact physical, emotional, social, cognitive, communications, worrying, daily activity and relationships in the family. It is scale with a scoring range from 0 to 4; a higher score indicates a better quality of life.
The PedsQL-Family Impact Module. | T2 (post-intervention in experimental group, 6 weeks after baseline).
  The Family Impact Module is an instrument of 37 items that measures family's quality of life. Eight sub-scales of parents functioning that compact physical, emotional, social, cognitive, communications, worrying, daily activity and relationships in the family. It is scale with a scoring range from 0 to 4; a higher score indicates a better quality of life.
Attention-deficit Hyperactivity Disorder Rating Scale - IV (ADHD-RS) | T1 (at baseline in experimental group).
  The ADHD-RS a checklist for children aged 5-17 years old for diagnosing ADHD in the classification found in the Diagnostic and Statistical Manual of Mental Disorder, 4th Edition (DSM-IV) and/or in the 10th revision of the International Statistical Classification of Diseases (ICD-10). The questionnaire has 18 items that consists of two subscales: in attention (9 items) and hyperactivity-impulsivity (9 items). Higher score indicates more symptoms.
Attention-deficit Hyperactivity Disorder Rating Scale - IV (ADHD-RS) | T2 (post-intervention in experimental group, 6 weeks after baseline).
  The ADHD-RS a checklist for children aged 5-17 years old for diagnosing ADHD in DSM-IV and ICD-10. The questionnaire has 18 items that consists of two sub-scales: in attention (9 items) and hyperactivity-impulsivity (9 items). Higher score indicates more symptoms.
Disruptive Behavior Rating Scale (DBRS) | T1 (at baseline in experimental group).
  The DBRS is an 8-statement rating-scale were parents list the symptoms of op-positional defiant disorder (ODD) and conduct disorder (CD). The scale is with a scoring range from 0 to 4; a higher score indicates more anti-developmental disorder.
Disruptive Behavior Rating Scale (DBRS) | T2 (post-intervention in experimental group, 6 weeks after baseline).
  The DBRS is an 8-statement rating-scale were parents list the symptoms of op-positional defiant disorder (ODD) and conduct disorder (CD). The scale is with a scoring range from 0 to 4; a higher score indicates more anti-developmental disorder.
Rosenberg Self-Esteem Scale | T1 (at baseline in experimental group).
  The Rosenberg Self-Esteem scale is a 10-item questionnaire for adolescents that measures self-worth by measuring both positive and negative feelings about the self-esteem. It is a 4-point scale format ranging from strongly agree to strongly disagree. Higher scores indicate higher self-esteem of positive thinking for building resilience.
Rosenberg Self-Esteem Scale | T2 (post-intervention in experimental group, 6 weeks after baseline).
  The Rosenberg Self-Esteem scale is a 10-item questionnaire for adolescents that measures self-worth by measuring both positive and negative feelings about the self-esteem. It is a 4-point scale format ranging from strongly agree to strongly disagree. Higher scores indicate higher self-esteem of positive thinking for building resilience.
Perlin´s Self-Mastery Scale | T1 (at baseline in experimental group).
  The Mastery scale is a 7-items questionnaire for adolescents. It is a 4-point scale format ranging from strongly agree to strongly disagree. A higher score indicates a better mastery.
Perlin´s Self-Mastery Scale | T2 (post-intervention in experimental group, 6 weeks after baseline).
  The Mastery scale is a 7-items questionnaire for adolescents. It is a 4-point scale format ranging from strongly agree to strongly disagree. A higher score indicates a better mastery.
Background for parents questionnaire | T1 (at baseline in experimental group).
  Questions about gender, age, education, work, family status, diagnoses, other psychological treatments. Mostly open-ended questions.
Background questionnaire for adolescents' | T1 (at baseline in experimental group).
  Questions about gender, age, school and work. Mostly open-ended questions.

CONTACTS AND LOCATIONS:
Overall Officials: Ása V Þórisdóttir, PhD, Study Director — University of Iceland
Locations (1):
- University of Iceland, Faculty of Nursing, Reykjavik, Iceland

IPD SHARING:
Plan to Share IPD: No